CLINICAL TRIAL: NCT02013999
Title: Mobile Game-based Virtual Reality Rehabilitation Program for Upper Limb Dysfunction After Ischemic Stroke
Brief Title: The Development of Upper Extremity Rehabilitation Program Using Virtual Reality for the Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1306/208-005
Record Dates: First submitted 2013-12-03; First posted 2013-12-17 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Upper Extremity Dysfunction After the Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Virtual reality program (Experimental): mobile device for virtual reality program
  Interventions: Other: Virtual reality program for upper extremity rehabilitation
- Control (Active Comparator): standard occupuational therapy
  Interventions: Other: standard occupational therapy

INTERVENTIONS:
Other: Virtual reality program for upper extremity rehabilitation
  Arms: Virtual reality program
Other: standard occupational therapy
  Arms: Control

SUMMARY:
Using the upper extremity rehabilitation program developed by virtual reality would help the recovery upper extremity function in patients with stroke.

DETAILED DESCRIPTION:
This randomized, double-blind, controlled trial included 24 patients with ischemic stroke. The intervention group received 30 min of conventional occupational therapy (OT) and 30 min of the mobile upper extremity rehabilitation program using a smartphone and a tablet PC (MoU-Rehab). The controls (n = 12) received conventional OT alone for 1 h per day. Rehabilitation consisted of 10 sessions of therapy, 5 days per week, for 2 weeks. The outcome measures (Fugl-Meyer Assessment of the upper extremity [FMA-UE], Brunnstr¨om stage [B-stage] for the arm and the hand, manual muscle testing [MMT], modified Barthel index [MBI], EuroQol-5 Dimension [EQ-5D], and Beck Depression Inventory [BDI]) were assessed at the beginning and end of treatment, and at 1 month. User satisfaction was evaluated by a qestionnaire.

ELIGIBILITY:
Inclusion Criteria:

* ischemic or hemorrhagic stroke confirmed by brain imaging study
* upper extremity dysfunction
* possible to use a simple device

Exclusion Criteria:

* delirium, confusion or other evidence related to the consciousness
* uncontrolled medical or surgical disease
* unable to command to the order due to severe cognitive impairment
* visual impairment
* unable to sit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11-24 (Actual); Study Completion 2014-11-24 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer upper extremity scale | baseline(just before beginning the treatment), at the end of the treatment for 2 weeks, 1 month later of the end of the treatment for 2 weeks
  for motor evaluation

SECONDARY OUTCOMES:
brunnström stage | baseline(just before beginning the treatment), at the end of the treatment for 2 weeks, 1 month later of the end of the treatment for 2 weeks
  for motor evaluation
Modified Barthel Index | baseline(just before beginning the treatment), at the end of the treatment for 2 weeks, 1 month later of the end of the treatment for 2 weeks
  for ADL independence
Medical Research Council (MRC) Scale for Muscle Strength | baseline(just before beginning the treatment), at the end of the treatment for 2 weeks, 1 month later of the end of the treatment for 2 weeks
  for motor evaluation
Euroqol(EQ)-5D | baseline(just before beginning the treatment), at the end of the treatment for 2 weeks, 1 month later of the end of the treatment for 2 weeks
  EQ-5D
Virtual reality kinematic data | everytime when the patient uses program (automatically all recorded)
  Automatically recorded
questionnaire | at the end of the treatment for 2 weeks
  for user satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, Ph.D, Principal Investigator — Seoul National University Bundang Hospital, Seongnam, South Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea